CLINICAL TRIAL: NCT03838458
Title: Comparison of Structural and Molecular Genetic Properties Between Normal and Hypospadic Children's Prepuces
Brief Title: Molecular and Structural Comparison of Hypospadic and Normal Children Prepuces
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Irem Inanc, MD, Trakya University
Other Study IDs: Hypospadic prepuce structure
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Hypospadias
Keywords: hypospadias; prepuce; HOXA13; FGFR2; TGF beta
MeSH Terms: conditions — Hypospadias; Camurati-Engelmann Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Preputial tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study: Children with isolated hypospadias
- Control: Children with planned circumcision

SUMMARY:
The aim of this study is to compare prepuce tissue samples from healthy male children who applied for circumcision and children with isolated hypospadias. Estrogen receptor 1 (ER1), androgen receptor (AR), FGFR2, transforming growth factor beta (TGF beta) and HOXA13 gene expression in the prepuce is planned to investigate via polymerase chain reaction (PCR) method. Mucosal vascular and nerve densities, and extracellular matrix density of laminin and collagen protein is planned to investigate via immunohistochemical examination.

ELIGIBILITY:
Inclusion Criteria:

* To apply for circumcision, not to have any genitourinary abnormalities/conditions for control group.
* To have isolated hypospadias for study group.

Exclusion Criteria:

* To have genitourinary surgery before.

Max Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: 0-18 years old pediatric male population, patients with isolated hypospadias are study group, patients with planned circumcision are control group.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Genetic analysis 1 | 1 year
  Androgen receptor (AR) gene PCR analysis
Genetic analysis 2 | 1 year
  Estrogen receptor 1 (ER1) gene PCR analysis
Genetic analysis 3 | 1 year
  FGFR2 gene PCR analysis
Genetic analysis 4 | 1 year
  TGF beta gene PCR analysis
Genetic analysis 5 | 1 year
  HOXA13 gene PCR analysis
Immunohistochemical study 1 | 1 year
  Mucosal vessel density is planned to determine via CD34
Immunohistochemical study 2 | 1 year
  Mucosal nerve density is planned to determine via PGP 9.5
Histological study 1 | 1 year
  Laminin is planned to determine in extracellular matrix via light microscope
Histological study 2 | 1 year
  Collagen is planned to determine in extracellular matrix via light microscope

CONTACTS AND LOCATIONS:
Overall Officials: Dincer Avlan, Profesor, MD, Principal Investigator — Trakya University Faculty of Medicine, Pediatric Surgery Department
Locations (1):
- Trakya University Faculty of Medicine, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided